CLINICAL TRIAL: NCT01161615
Title: A Randomized, Multi-Center, Double-Blind, Placebo-Controlled Phase III Trial to Evaluate the Efficacy, Tolerability and Safety of MRX-7EAT Etodolac-Lidocaine Topical Patch in the Treatment of Tendonitis and Bursitis of the Shoulder
Brief Title: MRX-7EAT Etodolac-Lidocaine Topical Patch in the Treatment of Tendonitis and Bursitis of the Shoulder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MEDRx USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRX-7EAT-1006
Record Dates: First submitted 2010-07-12; First posted 2010-07-13 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Acute Tendonitis; Bursitis
Keywords: tendonitis and/or bursitis of the shoulder; acute tendonitis and/or bursitis of the shoulder
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Therapy with placebo
  Interventions: Drug: Placebo
- MRX-7EAT (Experimental): Therapy with experimental drug
  Interventions: Drug: MRX-7EAT

INTERVENTIONS:
Drug: MRX-7EAT — Application of up to two patches for up to 7 days.
  Arms: MRX-7EAT
Drug: Placebo — Application of up to two patches for up to 7 days.
  Arms: Placebo

SUMMARY:
A Randomized, Multi-Center, Double-Blind, Placebo-Controlled Phase III Trial to Evaluate the Efficacy, Tolerability and Safety of MRX-7EAT Etodolac-Lidocaine Topical Patch in the Treatment of Tendonitis and Bursitis of the Shoulder.

ELIGIBILITY:
Main Inclusion Criteria:

* Subject is 14 years of age or older (with assent according to state law).
* Females of child bearing potential must have a negative pregnancy test.
* Subject has a diagnosis of acute tendonitis or bursitis of one shoulder with the onset of the current episode 5 days and ≤ 21 days preceding the screening visit. Diagnosis is indicated by a positive Hawkins Test and Neer Test, both resulting in pain with motion and the existence of shoulder impingement related to tendonitis or bursitis.
* Subject has a Current Pain Intensity rated prior to study entry ≥ 5 but ≤ 8 on a Numeric Pain Rating Scale (NPRS) (11 point; range 0 to 10; anchors to be "none" and "severe").

Main Exclusion Criteria:

* Subject has a suspected tear in the rotator cuff, calcific tendonitis.
* Standard of Care (SOC) diagnosis with an AP and lateral x-ray, adhesive capsulitis, shoulder fractures, bilateral tendonitis or bursitis of the shoulders; or orthopedic surgical treatment is required.
* Subject has a positive Drop Arm Test indicative of a suspected tear; a positive O'Brien's Test suggestive of a glenoid labral tear; a positive Apprehension Test which would be indicative of glenohumeral instability.
* Subject had a previous episode of shoulder pain in the same area within two months.
* Subject received passive physical therapy treatments (e.g., deep heat or ultrasound) for the tendonitis/bursitis for the target shoulder within the past 24 hours; requires continued use of an immobilization device for treatment of the current episode of tendonitis or bursitis or use of iontophoresis.
* Subject has used oral pharmacologic treatment (NSAIDs or analgesic medications) less than 3 half-lives before the baseline assessments; ibuprofen is permitted prior to baseline as long as it is not within 6 hours of the baseline assessment.
* Subject has used any form of opioid within 24 hours of study entry or use of opioids for 5 or more consecutive days within the 30 days preceding enrollment.
* Subject has received systemic corticosteroids in the 30 days preceding the screening visit.
* Subject recently initiated sleep medications, muscle relaxants, anticonvulsants or antidepressants.
* Subject used TNF alpha blockers or Class 1 anti-arrhythmic drugs within the past 60 days.
* Subject has a history or physical assessment finding of clinically significant.
* GI ulcers or abnormal bleeding, anemia, kidney disease, liver disease, poorly controlled lung, stomach, heart, or other vital organ disease as determined by the study investigator/physician.
* Subject has a history or physical assessment finding that is not compatible with safe participation in the study.
* Subject has a pain or medical problem that in the investigator's opinion may interfere with pain measurement of the target joint.
* Subject has active skin lesions or disease at the intended site of application of the study medication.
* Subject has a history of allergy to etodolac, other NSAIDs, lidocaine or adhesives (e.g., adhesive tape).
* Subject has a history of prior failed treatment with topical NSAIDs.
* Subject has a history of drug or alcohol abuse.
* Subject received an investigational drug within a period of 30 days prior to receiving study medication.
* Subject is scheduled for elective surgery or other invasive procedures during the period of study participation.
* Subject is on workman's compensation or has pending legal hearings.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2010-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Mean of all 24 Current Pain Intensity scores collected on Days 2 through 7 on a 0-10 NPRS. | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Martine Francis, Study Chair — IL Pharma
Locations (34):
- United States (34):
  - Chandler, Arizona
  - Phoenix, Arizona
  - North Little Rock, Arkansas
  - Chico, California
  - Mission Hills, California
  - Palm Springs, California
  - San Diego, California
  - Aurora, Colorado
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Daytona Beach, Florida
  - Fort Lauderdale, Florida
  - Gulf Breeze, Florida
  - Orlando, Florida
  - West Palm Beach, Florida
  - Avon, Indiana
  - Fishers, Indiana
  - Franklin, Indiana
  - Greenfield, Indiana
  - Muncie, Indiana
  - Dubuque, Iowa
  - Wichita, Kansas
  - Erlanger, Kentucky
  - Henderson, Nevada
  - Charlotte, North Carolina
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Georgetown, Texas
  - Lubbock, Texas
  - San Antonio, Texas
  - Temple, Texas
  - Riverton, Utah
  - Danville, Virginia